CLINICAL TRIAL: NCT06466876
Title: Retrieval-Based Word Learning in Autism Spectrum Disorder
Brief Title: Retrieval-Based Word Learning in Autistic Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Eileen Haebig, Associate Professor, Louisiana State University and A&M College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R21DC018872 (NIH); R21DC018872 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; word learning; retrieval practice; test effect
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Within participant design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Word Learning (Experimental): Each autistic child will be taught novel words in a behavioral task.
  Interventions: Behavioral: retrieval-based word learning

INTERVENTIONS:
Behavioral: retrieval-based word learning — Word learning intervention that compares two strategies for teaching novel words

SUMMARY:
Children on the autism spectrum sometimes have difficulty learning new words and using the newly taught information in different situations. In this study, the investigators are testing whether strategies that have been found to improve word learning in non-autistic children will also help autistic children. Specifically, the investigators aim to test whether autistic children learn words more successfully if novel words are taught by repeating the words to the child (re-study) or if the novel words are taught first with labeling each word and then quizzing the child (repeated quizzing).

The main questions it aims to answer are:

* When teaching nouns (names of exotic animals), is learning stronger if autistic children re-study or engage in repeated quizzing of the newly taught words?
* When teaching adjectives (visible features of objects, like a bumpy chair), is learning stronger if autistic children re-study or engage in repeated quizzing of the newly taught adjectives?
* Does the word learning condition (re-study vs. repeated quizzing) impact whether autistic children are more successful in demonstrating their knowledge of the newly taught words in different contexts?
* Are autistic features related to patterns of word learning?

Participants will:

* Learn new words with half of the words being taught in one way (re-study) and the other half of the words being taught in the other way (repeated quizzing).
* Participate in 5-minute and 1-week tests of the newly taught words to measure child learning.
* Complete other language, thinking, and autism clinical assessments.

DETAILED DESCRIPTION:
There is a rich literature in cognitive psychology that highlights the importance of opportunities to recall and produce newly taught information when learning. The use of retrieval practice during a learning phase improves long-term retention between 50% and 150% relative to conditions without retrieval prompts. Recent work documents the power of retrieval practice in word learning studies with preschoolers with developmental language disorders. Though retrieval practice is not new, its application to child learning is in its infancy. Given the striking learning effects that have been documented in adults and emerging findings in children [with language impairment, retrieval practice has great potential to enhance learning in autistic children, a population with significant vocabulary deficits that often persist into adulthood.

Though autistic children have initial strengths in learning word form information (phonological), these word form advantages do not persist over time. Autistic children also demonstrate weaknesses in developing robust semantic representations, which have been noted by recalling fewer semantic features of newly taught words. Also, autistic children have difficulties in generalizing newly taught knowledge, which can hinder flexible vocabulary use. It has been suggested that autistic children may need more input, time, or practice than typically developing children to develop strong lexical representations.

In addition to deficits in breadth and depth of word knowledge, many autistic children demonstrate an atypical receptive-expressive vocabulary profile, with a reduced receptive advantage. Despite traditional therapy approaches recommending that receptive skills be targeted before expressive skills in autistic children, research indicates that it may be more effective to target expressive skills (i.e., word production) prior to targeting receptive skills. One recent study demonstrated that autistic children are more successful when learning words if they are prompted to name newly taught items rather than to identify (point to) a picture of these items. Targeting word expression led to more successful cross-modal generalization, with success extending to word comprehension (i.e., expressive-to-receptive generalization). This new finding holds promise for clinical practice; however, it has not been connected to a strong mechanistic explanation, which is necessary to strengthen the support for this practice. Retrieval-practice theory can provide the key mechanistic explanation that is required.

It has been proposed that effortful retrieval (now referred to as repeated spaced retrieval; RSR for clarity) enhances encoding because the retrieval of new information, or the attempt to do so, prompts individuals to identify features of the word or concept that are necessary to reconstruct the material, which leads to the development of an enriched and potentially elaborated memory trace to support future retrievals. RSR holds promise for autistic children because it may strengthen item-specific learning of phonological and semantic information (word form and meaning) that persists beyond immediate tests of learning. Furthermore, RSR may enable generalization (e.g., applying noun labels to new referents and adjectives to different objects). Thus, our specific aims are:

Aim 1: To determine whether repeated spaced retrieval (RSR) of labels (nouns) results in more robust learning of word form and meaning relative to a learning schedule that does not prompt retrieval.

In Study 1, 4- to 10-year-old autistic children will learn [novel nouns] in an RSR condition and a Repeated Study only (RS) condition. The investigators hypothesize that the children will recall more labels (word form) and semantic information (meaning) for RSR words and that their learning gains will persist at the 1-week test.

Aim 2: To determine whether repeated spaced retrieval (RSR) of adjectives results in more robust learning relative to a learning schedule that does not prompt retrieval. Study 2 will examine novel adjective learning, which has not been examined in autistic children. Autistic children will learn novel adjectives for unusual attributes displayed on familiar objects (e.g., "The cow is zogy."). It is predicted that the children will benefit from the RSR schedule when learning adjectives at immediate and 1-week tests.

Aim 3: To determine whether RSR enhances learning to the extent that children are able to generalize newly learned words to new images/referents. To demonstrate durable learning, the investigators will test beyond the explicitly taught stimuli. Study 1 will examine whether children will extend the labels (nouns) to referents that differ slightly in positioning and color. Study 2 will test for generalization of the newly taught adjectives when applied to objects from different categories (e.g., a zogy cow [taught] and zogy table [generalization]). It is predicted that generalization will be higher for words taught in the RSR condition than the RS condition.

Aim 4: To explore the moderating effect of autism severity on response to RSR. The investigators will examine whether autism symptom severity moderates word learning overall and if it predicts whether children benefit from RSR relative to RS learning schedules in Studies 1 and 2. The investigators will also explore associations between word learning and cognitive, vocabulary, and grammatical skills, and when warranted, statistically control for these variables.

ELIGIBILITY:
Inclusion Criteria:

* Children with autism spectrum disorder (ASD) will participate in this study. The study will be 4- to 10-years-old and will already have a community diagnosis of autism spectrum disorder. The diagnosis will be confirmed confirmed using the Autism Diagnostic Observation Schedule - 2nd edition (ADOS-2; Lord et al., 2012).
* Because the children will be completing an experimental word learning study that requires the child to verbally produce the newly taught words, children must have verbal communication skills (i.e., be able to speak in at least simple sentences spontaneously), which will be determined in initial correspondence with the child's parent or guardian.
* Children's primary language spoken must be English.
* All children will pass a hearing screening.
* Additionally, all children will score above 75 on the Leiter-3 (Roid, Miller, & Pomplun, 2013), a nonverbal cognitive assessment.

Exclusion Criteria:

* Because the word learning study involves the child needing to produce the taught words non-speaking autistic children and minimally speaking autistic children (i.e., is not able to produce at least simple sentences in spontaneous speech) will be excluded from the proposed studies.
* If the child has a history of a neurological disorder such as cerebral palsy or a known genetic disorder that causes developmental delays/disorders
* If the child has an un-corrected hearing loss.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Word form recall | During the 5-minute test and 1-week test (for taught and generalization referents) for Studies 1 and 2
  For Study 1 and 2, we will document child learning with higher scores indicating better learning.
  Measures: Accuracy -- overall accuracy assigning 0-1 points for each word (minimum: 0, maximum: 16) and phonological accuracy assigning multiple points based off of the adapted scoring procedures from Edwards et al. (2004).
Word meaning recall | During the 5-minute test and 1-week test (for taught and generalization referents) for Studies 1 and 2
  For Study 1 (noun learning), we will document child learning with 0 and 1 values that will be summed across test items. Higher scores indicating better learning Word meaning will be assessed by asking children to recall/state: 1) what each animal likes and 2) what each animal likes to do.
  Measure: Accuracy -- overall accuracy assigning 0 - 1 point for each word meaning that is accurately recalled (likes meaning score minimum: 0, maximum: 16, likes to do meaning score minimum: 0, maximum: 16)
Form-referent-link recognition | During the 1-week test (for taught and generalization referents) for Studies 1 and 2
  For Study 1 and 2 at the 1-week test, we will test children's receptive knowledge of the newly taught words (nouns and adjectives) and their ability to demonstrate generalization. The form-referent link recognition tests will be a multiple-choice measure in which the child is asked to point to the referent in an array consisting of the target and two foils. The foils will be picture referents of the other novel words in the study. Measure: Accuracy -- 0 - 1 point for each accurate response Minimum: 0, Maximum: 16 Higher scores indicate better learning.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen K Haebig, PhD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Louisiana State University, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data will be shared on national databases (e.g., NDAR) or with collaborators, we will only do so for participants whose parents who have explicitly provided permission on the consent form to have their data shared with other researchers for future related studies.

REFERENCES:
- [Background] Leonard LB, Karpicke J, Deevy P, Weber C, Christ S, Haebig E, Souto S, Kueser JB, Krok W. Retrieval-Based Word Learning in Young Typically Developing Children and Children With Developmental Language Disorder I: The Benefits of Repeated Retrieval. J Speech Lang Hear Res. 2019 Apr 15;62(4):932-943. doi: 10.1044/2018_JSLHR-L-18-0070. PMID 30986142